CLINICAL TRIAL: NCT05195879
Title: A Phase I Study to Evaluate Safety, Biodistribution, Radiation Dosimetry, and Pharmacokinetics of XTR004 in Healthy Chinese Volunteers
Brief Title: A Study of XTR004 Radiotracer in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sinotau Pharmaceutical Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STB-XTR004-101
Record Dates: First submitted 2021-07-22; First posted 2022-01-19 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Coronary Artery Disease (CAD); Myocardial Ischemia
Keywords: coronary artery disease; positron emission tomography; myocardial perfusion imaging; XTR004
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XTR004 (Experimental): Single dose 6.0-8.0 mCi intravenous injection of XTR004 and investigation of XTR004 (MPI radiotracer).
  Interventions: Diagnostic Test: XTR004

INTERVENTIONS:
Diagnostic Test: XTR004 — Single dose intravenous injection of XTR004. Serial whole-body PET scan will be obtain after injection, blood and urine collection after injection for the assessment of pharmacokinetics.

SUMMARY:
XTR004 is a 18F-labeled myocardial perfusion positron emission tomography tracer use to measure myocardial perfusion and myocardial blood flow. XTR004 binds to the myocytes and targets respiratory chain complex 1 in the mitochondria.This phase I study investigated the safety, biodistribution, radiation dosimetry and Pharmacokinetics of XTR004 in 10 healthy Chinese adults volunteers.

DETAILED DESCRIPTION:
XTR004 is a 18F-labeled myocardial perfusion PET tracer, the first one developed in China by Sinotau Pharmaceutical Group. XTR004 targets and binds to the mitochondrial complex I protein. XTR004 reflects myocardial function at a molecular level. In pre-clinical studies XTR004 demonstrated high myocardial first-pass extraction and prolonged retention, allowing for early or delayed imaging. XTR004 can be clinically used to measure myocardial perfusion and myocardial blood flow. This Phase I study will be open-labeled, nonrandomized, single center study. Enrolled 10 healthy Chinese adults who meet all of the inclusion and none of the exclusion criteria. Subjects will receive 6-8 mCi of XTR004 via IV injection. Safety and tolerability will be observed. Biodistribution, pharmacokinetics, and dosimetry will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese men and women are included age between 18-40 years
2. Normal vital signs and physical examination
3. No clinical abnormalities in ECG, EEG, and echocardiogram
4. No past history of cardiovascular, cerebrovascular, or gastrointestinal diseases
5. Normal or no clinical significance abnormalities in laboratory tests
6. No any other major or chronic illness
7. No presence of drug use
8. Females adopt effective medically approved contraceptive methods to prevent pregnancy for at least 6 months before the study and after the study
9. Voluntarily agree and signed written consent

Exclusion Criteria:

1. Previous history of cardiovascular diseases
2. A history of or physical or radiographic manifestations of any previous brain disease
3. Any previous major disease or unstable condition
4. Subjects who cannot complete XTR004 imaging as required
5. Positive HIV, hepatitis C or Treponema pallidum antibody and hepatitis B surface antigen detection
6. A history of coagulation or coagulation disorder
7. A history of liver or gastrointestinal disease or other conditions that interfere with drug absorption, distribution, excretion or metabolism as determined by the investigator
8. Previous history of cancer
9. High risk of drug allergic reaction
10. A history of alcohol or drug abuse/dependence
11. Exposure to significant occupational radiation (e.g >50 mvs/year) or exposure to radioactive substances for therapeutic or research purposes over the past 10 years
12. Scheduled surgery or other invasive interventions within one week before drug injection
13. Subjects use any drug or treatment that may interfere with the experimental data or cause serious side effects, as determined by the investigator
14. Pregnant or lactating women
15. Admitted to hospital due to illness during screening period Other conditions that investigators consider inappropriate to participate in a trial.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Physical examination of the major organ systems | up to 14 days post injection
  Safety observation: Observation of Cardiovascular system (blood pressure, pulse rate, and rhythm), Lungs (respiratory rate, chest expansion, and lung auscultation), Abdominal system (for any tenderness or organ enlargement), Nervous system ( cognitive testing, motor strength and control, including mental status), Musculoskeletal system, and Skin for any abnormalities, after drug injection. To report number of participants with changes in physical examination compared to baseline physical examination obtained before drug injection.
12-lead Electrocardiography | up to 14 days post injection
  Safety observation: Observation of ECG electrical activity pattern in the P-wave, PR interval, QRS wave complex, ST segment, and T-wave if associated with any abnormality after drug injection. To observe and report participants with ECG abnormality compared to baseline ECG obtained before drug injection.
Monitoring of body temperature | up to 14 days post injection
  Safety observation: Vital sign monitoring of body temperature (degrees celsius ) after drug injection. To report changes in body temperature compared to baseline body temperature obtained before drug injection.
Monitoring of respiratory rate | up to 14 days post injection
  Safety Observation: Vital sign monitoring of respiratory rate (breath per minute) after drug injection. To report changes in respiratory rate compared to baseline respiratory rate obtained before drug injection.
Monitoring of Blood pressure | up to 14 days post injection
  Safety Observation: Vital sign monitoring of blood pressure (mmHg) after drug injection. To report changes in blood pressure compared to baseline blood pressure obtained before drug injection.
Monitoring of pulse rate | up to 14 days post injection
  Safety Observation: Vital sign monitoring of pulse rate (beats per minute) after drug injection. To report changes in pulse rate compared to baseline pulse rate obtained before drug injection.
Changes in Laboratory tests | up to 14 days post injection
  Safety observation: Measurements of routine blood (g/L), routine urine (mg/dL), and blood troponin-I levels (ng/ml) after drug injection. To observe and report changes in routine blood, routine urine, and blood troponin-I levels compared to baseline values obtained before drug injection.
Incidence of adverse events | up to 14 days post injection
  Safety Observation: Number of participants with adverse events and severe adverse events after drug injection.

SECONDARY OUTCOMES:
Biodistribution of XTR004 after a single dose IV injection. PET scan acquisition; | up to 4.5 hours
  Whole-body PET scan obtained at the following time points; at 0-60, 120, 150, 240, and 270 minutes, post injection.
Plasma and blood radioactivity analysis | up to 7 hours
  Venous blood collection of 6ml at 1.5, 3, 5, 10, 30, 60, 120, 240 and 420 minutes for plasma and blood radioactivity analysis, post injection
Urine radioactivity analysis | up to 7.25 hours
  Urine will be collected up to ~ 7.25 hours to assess for radioactivity, post injection.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No